CLINICAL TRIAL: NCT04106908
Title: MOdalities of Use, effectiveNEss and TOlerability of Eqwilate® a Balanced combInatiON of VWF and FVIII in Von WillEbrand Patients in Real-life Conditions: the ONE-TO-ONE Study
Brief Title: Effectiveness and Tolerability of Eqwilate in Real-life Conditions
Status: Active, not recruiting | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: WIL-32
Record Dates: First submitted 2019-08-28; First posted 2019-09-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: VWD - Von Willebrand's Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eqwilate
  Interventions: Biological: Eqwilate

INTERVENTIONS:
Biological: Eqwilate — Eqwilate® is a new generation, albumin-free, high-purity, double virus-inactivated, freezedried concentrate of VWF and FVIII

SUMMARY:
MOdalities of use, effectiveNEss and TOlerability of Eqwilate® a balanced combInatiON of VWF and FVIII in von WillEbrand patients in real-life conditions: the ONE-TO-ONE study

ELIGIBILITY:
Inclusion Criteria:

The study will involve patients (≥ 6 years of age) from the participating centres treated with Eqwilate® (either on-demand, as perioperative prophylaxis, or as prophylaxis) during the time inclusion period will be opened. Patients will be of any VWD type, previously treated or untreated.

Exclusion Criteria:

* N/A

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will involve patients (≥ 6 years of age) from the participating centres treated with Eqwilate® (either on-demand, as perioperative prophylaxis, or as prophylaxis) during the time inclusion period will be opened.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Haemostatic Effectiveness of On-demand Treatment | 12 months
  Haemostatic Effectiveness of On-demand Treatment (excellent, good, moderate, none)
  none: severe uncontrolled bleeding or intensity of bleeding not changed (in case of non-severe bleeding episodes); moderate: moderate bleeding, or control of bleeding required additional product; good: slight oozing and adequate control of bleeding episode and did not require additional product; excellent: haemostasis achieved, cessation of bleeding episode.
Haemostatic Effectiveness of Perioperative Prophylaxis | 12 months
  Haemostatic Effectiveness of Perioperative Prophylaxis (excellent, good, moderate, none)
  none: severe uncontrolled bleeding or intensity of bleeding not changed (in case of non-severe bleeding episodes); moderate: moderate bleeding, or control of bleeding required additional product; good: slight oozing and adequate control of bleeding episode and did not require additional product; excellent: haemostasis achieved, cessation of bleeding episode.
Occurrence of Bleeding Episodes During Follow-Up | 12 months
  Occurrence of Bleeding Episodes During Follow-Up

SECONDARY OUTCOMES:
FVIII Levels | 12 months
  Clotting factor VII levels in blood
Productivity Loss | 12 months
  Days lost from school or work
Volume of Blood loss | up to 1 week
  Volume of Blood loss
Immunogenicity Presence of inhibitors against VWF | 12 months
  Presence of inhibitors against VWF found via blood draw analysis

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Caen Study Site, Caen
  - Clamart Study Site, Clamart
  - Paris Study Site - Lariboisiere, Paris
  - Paris Study Site - Necker, Paris
  - Rennes Study Site, Rennes
  - Rouen Study Site, Rouen
  - Saint Denis Study Site - Pediatrie, Saint-Denis
  - Saint Denis Study Site, Saint-Denis
  - Saint-Etienne Study Site, Saint-Etienne